CLINICAL TRIAL: NCT01321996
Title: Employment of 68Ga-DOTA-NOC in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: 68Ga-DOTA-NOC PET/CT in Patients With Idiopathic Pulmonary Fibrosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: enrollment failure (only 29 patients were enrolled during the study period)
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Stefano Fanti, Associate Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CE119/2008/0/Sper
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: PET/CT; 68Ga-DOTANOC; IPF; NSIP; Idiopathic pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-DOTANOC PET/CT in patients with IPF and NSIP (Other): one arm study: all patients were studied by 68Ga-DOTANOC PET/CT
  Interventions: Procedure: 68Ga-DOTA-NOC PET/CT

INTERVENTIONS:
Procedure: 68Ga-DOTA-NOC PET/CT — procedure: PET/CT scan with 68Ga-DOTA-NOC

SUMMARY:
The investigators aim to evaluate the role of 68Ga-DOTA-NOC PET/CT in patients with idiopathic pulmonary fibrosis, in particular in patients with a diagnosis of IPF/UIP (idiopathic pulmonary fibrosis, diagnosed based in the American Thoracic Society and European Respiratory Society criteria) and in forms of NSIP (non-specific interstitial pneumonia). PET/CT imaging data will be compared with HRCT (high-resolution computed tomography) findings to assess disease extension, early disease detection and to non-invasively detect somatostatin receptors expression at lung level in these patients, with potential therapeutic implications.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis prognosis remains severe, in particular for IPF, the most common entity. Moreover, current treatment options are largely ineffective and do not change the natural course of the disease. Pre-clinical evidence supports somatostatin receptors expression in the lung of patients with IPF. Recently new PET tracers (Somatostatin analogues labelled with 68Gallium), specifically binding to somatostatin receptors, have been developed and are used in neuroendocrine tumours clinical trials.

Aim of the present study is to evaluate the role of 68Ga-DOTA-NOC PET/CT in patients with idiopathic pulmonary fibrosis, in particular in patients with IPF/UIP and in cases with NSIP, that are characterized by a more indolent progression. PET/CT data will be compared with HRCT findings for the early detection of fibrotic areas and to non-invasively assess somatostatin receptors expression at lung level in these patients, with potential therapeutic implications. Moreover, the SUVmax (maximum standardized uptake value) will be analyzed in comparison with disease site and extension on HRCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of IPF and NSIP, based on the American Thoracic Society/European Respiratory Society Consensus Conference
* age ≥ 18 years
* males/females
* signed informed consent

Exclusion Criteria:

* pregnancy
* breast feeding
* healthy volunteers
* paediatric cases
* patients in emergency situations
* patients legally incompetent
* patients who refuse to sign the informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Describe pattern of 68Ga-DOTA-NOC uptake in comparison with HRCT findings | timeframe between imaging procedures 30 days

SECONDARY OUTCOMES:
68Ga-DOTA-NOC SUVmax correlation with pulmonary function tests | timeframe between PET/CT and pulmonary fucntion tests 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Fanti, Professor, Principal Investigator — Nuclear Medicine, Azienda Ospedaliero Universitaria di Bologna, Policlinico S.Orsola Malpighi, Bologna, Italy
Locations (1):
- Nuclear Medicine, Azienda Ospedaliero Universitaria di Bologna, Policlinico S.Orsola Malpighi, Bologna, Italy

REFERENCES:
- [Result] Ambrosini V, Zompatori M, De Luca F, Antonia D, Allegri V, Nanni C, Malvi D, Tonveronachi E, Fasano L, Fabbri M, Fanti S. 68Ga-DOTANOC PET/CT allows somatostatin receptor imaging in idiopathic pulmonary fibrosis: preliminary results. J Nucl Med. 2010 Dec;51(12):1950-5. doi: 10.2967/jnumed.110.079962. Epub 2010 Nov 15. PMID 21078794